CLINICAL TRIAL: NCT06523738
Title: Association of Left Atrial Volume Changes After Cardioversion and Recurrence of Atrial Fibrillation After Radiofrequency Ablation in Patients With Persistent Atrial Fibrillation
Brief Title: Left Atrial Volume Changes Who Underwent Cardioversion and Recurrence of AF After RF Ablation in Persistent AF (SAFE-AF)
Acronym: SAFE-AF-ABL
Status: Recruiting | Type: Observational
Sponsor: The Second Affiliated Hospital of Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Yuehui Yin, Chief Director, The Second Affiliated Hospital of Chongqing Medical University
Other Study IDs: SAFE-AF-ABL
Record Dates: First submitted 2024-07-23; First posted 2024-07-26 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-07

CONDITIONS: Persisent Atrial Fibrillation; Reversal of Atrial Enlargement; Recurrence of Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Reversible Group: Left atrial volume (LAV) decreased by 15% 3 to 6 months after electrical/pharmacological cardioversion compared to baseline. Consequently, patients in the group will receive pulmonary vein isolation only.
  Interventions: Diagnostic Test: 1. electrical/pharmacological cardioversion. 2.pulmonary vein isolation
- Irreversible Group: Left atrial volume (LAV) decreased by less than 15% 3 to 6 months after electrical/pharmacological cardioversion compared to baseline. Patients in the group will receive pulmonary vein isolation only.
  Interventions: Diagnostic Test: 1. electrical/pharmacological cardioversion. 2.pulmonary vein isolation

INTERVENTIONS:
Diagnostic Test: 1. electrical/pharmacological cardioversion. 2.pulmonary vein isolation — 1. electrical/pharmacological cardioversion. 2. pulmonary vein isolation for persistent atrial fibrillation

SUMMARY:
Electrical/pharmacological cardioversion improves structural remodeling of left atrium. We hypothesize that persistent atrial fibrillation (AF) patients with more significant left atrial size reduction after cardioversion have lower AF recurrence rates following radiofrequency ablation. The aim is to evaluate the relationship between changes in left atrial size 3 to 6 months after cardioversion and the recurrence rate of atrial fibrillation following radiofrequency ablation.

DETAILED DESCRIPTION:
Background: Atrial fibrillation (AF) is estimated to affect over 33 million people worldwide and is associated with significant co-morbidities such as embolic stroke, heart failure, dementia. Consequently, AF poses a significant burden to the healthcare system, in both direct and indirect costs. The management of AF is complex, especially for patients with persistent AF, which is defined as sustained AF for > 7 days. It is preferable to terminate the AF and restore normal sinus rhythm for relief of symptoms associated with AF or improvement of cardiac structure and function. The maintenance of AF, especially persistent AF is associated with fibrosis of left atria. Furthermore, AF itself promotes fibrosis, which in turn leads to increased conduction heterogeneity within the atrial substrate resulting in further progression of AF. In animal models, alterations in myocytes after sustained AF resemble those of myocardial hibernation. Ultimately, these structural changes would lead to Calcium overload and metabolic stress, similar changes have been observed in humans. In humans, atrial dilatation and degenerative changes have been observed. Interstitial fibrosis is the prime cause of structural remodeling in left atrium. In AF patients who did not experience AF recurrence after catheter ablation, the reduction in left atrial size was more significant. In the past, a 15% reduction in left atrial volume has been defined as left atrial reverse remodeling and is associated with the maintenance of sinus rhythm after AF ablation. It remains unclear whether the reduction in left atrial size after the restoration of sinus rhythm through electrical or pharmacological cardioversion in patients with persistent AF can predict AF recurrence following radiofrequency ablation.

Objectives: To evaluate the relationship between changes in left atrial size 3-6 months after electrical or pharmacological cardioversion in patients with persistent AF and AF recurrence within one year following radiofrequency ablation.

Methods: This study will be an observational trial of patients with persistent AF. Candidates will be identified among inpatients or outpatients if they have had at least two echocardiograms, one before and one 3-6 months after pharmacological or electrical cardioversion. Heart rhythm will be assessed through medical records and telephone surveys.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with estabolished diagnosis of Persistent Atrial Fibrillation during past 6 mnths.
2. LAD brfore entering the two cohorts is more than 40mm, and less than 50mm.
3. Pharmacological or electrical cardioversion has be performed successfully.
4. At least two echocardiograms were performed before and 3-6 months after cardioversion., and confirm the status of LAD (Reversal, unchange, enlargment).
5. Patients have given informed consent.

Exclusion Criteria:

1. Prior radiofrequency ablation treatment for atrial fibrillation
2. Prior cardiac surgical procedures
3. Individuals with cognitive impairments who are unable to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Persistent atrial fibrillation patients with enlarged left atrium.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-07-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Recurrence of atrial fibrillation | 1, 3, 5 years
  Recurrence of atrial fibrillation after radiofrequency ablation

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided